CLINICAL TRIAL: NCT04621786
Title: Electroconvulsive Therapy Amplitude Titration for Improved Clinical Outcomes in Late Life Depression
Brief Title: Electroconvulsive Therapy Amplitude Titration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: The Zucker Hillside Hospital (Other); National Institute of Mental Health (NIMH) (NIH); The Mind Research Network (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MH125126; MH125126 (Other Grant/Funding Number: NIMH)
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Major Depressive Disorder
Keywords: Electroconvulsive Therapy; Depressive Episode; Cognition
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Masking Description: Subject and outcomes assessor were blinded to amplitude titration
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental arm (Experimental): All subjects enrolled will receive amplitude titration for their first treatment. The remainder of the ECT series will be completed with traditional (800mA) pulse amplitude with right unilateral electrode placement. This investigation only includes the single open-label arm.
  Interventions: Device: Mecta Spectrum 5000Q paired with Soterix Medical 4X1 HD - ECT Multi-Channel Stimulation Interface

INTERVENTIONS:
Device: Mecta Spectrum 5000Q paired with Soterix Medical 4X1 HD - ECT Multi-Channel Stimulation Interface — The Mecta Spectrum 5000Q paired with Soterix Medical 4X1 HD-ECT Multi-Channel Stimulation Interface will reduce ECT current amplitude for amplitude-seizure titration.

SUMMARY:
This study is focused on advancing ECT treatment for older adults with depressive disorders by refining neuromodulation stimulus parameters to improve efficacy and cognitive safety.

DETAILED DESCRIPTION:
Amplitude titration, as proposed in this current proposal, can reduce the variability related to fixed amplitude dosing and optimize clinical and cognitive outcomes. The goal of this project is to change standard ECT parameter selection from a fixed amplitude to an individualized and empirically determined amplitude. To achieve this goal, the investigators will focus on the relationship between amplitude titration and treatment-responsive changes in hippocampal neuroplasticity with RUL fixed amplitude ECT. Fixed amplitude ECT results in variable E-field or ECT dose. Over the course of an ECT series, the variable ECT dose will result in inconsistent changes in hippocampal neuroplasticity. In contrast, pre-translational investigations have demonstrated that amplitude titration results in a consistent E-field or ECT "dose". Seizure titration amplitudes (based on historic data, 233 to544mA) are below the amplitude range of FDA-approved ECT devices (500 to 900mA) and will require an adaptor to reduce the output amplitude (Investigational Device Exemption). Amplitude titration will also be below the hippocampal neuroplasticity threshold and insufficient for antidepressant response. The difference between RUL amplitude titration and RUL fixed amplitude (800mA) ECT will determine the degree of target engagement with the hippocampus. To illustrate, subjects with low amplitude titration of ~250 mA (800/250, high fixed/titration amplitude ratio) will have significant changes in hippocampal neuroplasticity. Subjects with high amplitude titration ~500mA (800/500, low fixed/titration ratio) will have minimal changes in hippocampal neuroplasticity. The relationship between amplitude titration and fixed amplitude hippocampal neuroplasticity will be used to develop the amplitude multiplier required for consistent and clinically effective ECT dosing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder
* Clinical indications for ECT with right unilateral electrode placement
* Right-handed
* Age range between 50 and 80 years

Exclusion Criteria:

* Defined neurological or neurodegenerative disorder (e.g., traumatic brain injury, epilepsy, Alzheimer's disease)
* Other psychiatric conditions (e.g., schizophrenia, bipolar disorder)
* Current drug or alcohol use disorder (except for nicotine); and 4) contraindications to MRI.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental Arm
Started | 41
Completed | 29
Not Completed | 12
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Amplitude determined seizure [Mean (Standard Deviation); unit: milliamperes] — The first treatment used a method of limits to determine the amplitude (milliamperes) necessary to induce seizure activity.
  milliamperes | 312 (113)

OUTCOME MEASURES:

1. Primary Outcome: Beta Coefficient From Linear Regression of Amplitude-determined Seizure (Independent Variable) and Ebrain (Dependent Variable)
Description: Electric field modeling is used to calculate Ebrain from the pre-ECT structural MRI. Ebrain is an individual's electric field strength (Volts/meter) per unit current (milliampere). To avoid confounds from the tissue boundary effects, Ebrain is calculated as the 90th percentile of maximal. Higher values (0.2 Volts/meter per milliampere) indicate that an individual receives a higher electric field strength per unit current. The Ebrain in this sample ranges from 0.1 to 0.19 Volts/meter per milliampere. Linear regression model assessed the relationship between amplitude-determined seizure (independent variable) and Ebrain (dependent variable) with beta coefficient and 95% confidence intervals.
Time Frame: First treatment
Population: Amplitude determined seizure (miliamperes) predicting Ebrain (Volts/meter per milliampere)
Measure: Least Squares Mean (95% Confidence Interval); unit: beta coefficient from linear regression
Arm/Group | Experimental Arm
Number analyzed (Participants) | 29
beta coefficient from linear regression | -.0001054 [-.0001767 to -.0000341]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 0/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=29)
Attempted self-harm (Psychiatric disorders) | 1 (1) — Subject attempted self-harm and was hospitalized during protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT04621786/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/86/NCT04621786/SAP_003.pdf